CLINICAL TRIAL: NCT02391363
Title: Calmer Life: Treating Worry Among Older Adults In Underserved, Low-income, Minority Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Melinda Stanley, Professor and Head, Division of Psychology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AD-1310-06824
Record Dates: First submitted 2015-02-26; First posted 2015-03-18 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-02

CONDITIONS: Anxiety
Keywords: anxiety; worry
MeSH Terms: conditions — Anxiety Disorders | interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calmer Life (Experimental): Cognitive behavior treatment for anxiety
  Interventions: Behavioral: Cognitive behavior treatment
- Enhanced Community Care (Active Comparator): Enhanced information and referral services for mental health and basic needs
  Interventions: Behavioral: Information and referral

INTERVENTIONS:
Behavioral: Cognitive behavior treatment — Anxiety management skills with the option to included religious/spiritual beliefs and practices
  Arms: Calmer Life
Behavioral: Information and referral — Resource counseling and follow-up for mental health and basic needs
  Arms: Enhanced Community Care

SUMMARY:
The purpose of this research study is to see how helpful two different interventions offered through the Calmer Life program are in reducing worry and improving mood. The investigators also want to understand how a program like Calmer Life can be offered in underserved communities.

DETAILED DESCRIPTION:
Background: Recurrent, excessive, uncontrollable worry about multiple topics is common in older adults, but it is not well studied. This significant worry can negatively affect thinking, and it is associated with poorer sleep, more depression, and worse general health. Despite its prevalence, researchers have not studied significant worry enough, particularly in low-income racial and ethnic minority populations. We know these groups are unlikely to have adequate mental health care. We also know that older adults and minorities prefer treatments for worry that do not require medication, and that these kinds of treatments can be effective. Additional tests of treatments that do not involve drugs are needed in low-income racial and ethnic minority populations. Such person-centered research could expand access to appropriate care.

Objectives: The study team plans to compare two approaches, one called Calmer Life (CL) and another called Enhanced Community Care (ECC). CL helps individuals by providing worry-reduction skills and resource counseling for basic needs in a flexible, culturally supportive manner. ECC relies on standard information and resource counseling. The study will answer three questions. First, compared to ECC, is CL more effective at relieving significant worry? Second, which one is more effective at reducing anxiety and depression and improving sleep, ability to do daily activities, and use of medical services? Third, are improvements still present three months after treatment concludes?

Methods: In agreement with our community partners and governed by a council of community leaders, consumers, and providers from low-income minority communities, we will conduct the study. This community-academic partnership, created four years ago, introduced CL to the community. Case managers and community health workers from partner organizations were trained to implement CL. They taught worry-reduction skills and helped participants increase their use of community resources. Content was flexible so that participants could choose which skills to learn and whether or not to include religion or spirituality. They also could learn skills at home, by telephone, or in the community. In a new, larger comparison study, we will enroll 120 women and 30 men who are 50 years of age or older with significant worry. Most (80 percent) will be African American, and 70 percent will have income below poverty. Participants will be assigned by chance to CL or ECC and treated for six months. Brief assessments at enrollment and at six and nine months will rely on participants' reports. Differences will be measured statistically.

ELIGIBILITY:
Inclusion Criteria:

* PSWQ greater than 22

Exclusion Criteria:

* PHQ score less than 20
* Active suicidal intent
* Active psychosis or bipolar disorder
* Substance abuse
* Cognitive impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2014-11; Primary Completion 2017-09 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda A Stanley, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- VA HSR&D Center for Innovations in Quality, Effectiveness & Safety (IQuESt), Houston, Texas, United States

REFERENCES:
- [Derived] Stanley MA, Wilson NL, Shrestha S, Amspoker AB, Wagener P, Bavineau J, Turner M, Fletcher TL, Freshour J, Kraus-Schuman C, Kunik ME. Community-Based Outreach and Treatment for Underserved Older Adults With Clinically Significant Worry: A Randomized Controlled Trial. Am J Geriatr Psychiatry. 2018 Nov;26(11):1147-1162. doi: 10.1016/j.jagp.2018.07.011. Epub 2018 Aug 7. PMID 30224269
- [Derived] Steiner AJ, Boulos N, Wright SM, Mirocha J, Smith K, Lopez E, Gohar SH, Ishak WW. Major Depressive Disorder in Patients With Doctoral Degrees: Patient-reported Depressive Symptom Severity, Functioning, and Quality of Life Before and After Initial Treatment in the STAR*D Study. J Psychiatr Pract. 2017 Sep;23(5):328-341. doi: 10.1097/PRA.0000000000000251. PMID 28961662
- [Derived] Shrestha S, Wilson N, Kunik ME, Wagener P, Amspoker AB, Barrera T, Freshour J, Kraus-Schuman C, Bavineau J, Turner M, Stanley MA. Calmer Life: A Hybrid Effectiveness-implementation Trial for Late-life Anxiety Conducted in Low-income, Mental Health-Underserved Communities. J Psychiatr Pract. 2017 May;23(3):180-190. doi: 10.1097/PRA.0000000000000234. PMID 28492456

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from February 2015 through October 2016 in community settings where older adults gather and/or receive services such as social service agencies, churches, senior housing and community centers.
Pre-assignment Details: Prior to random assignment, participants were screened at three separate times. During this process, 84 participants were ineligible due to presence of exclusionary criteria, 24 were lost to follow-up and 5 withdrew from the study.
Period: Overall Study
Arm/Group | Calmer Life | Enhanced Community Care
Started | 70 | 64
Completed | 59 | 56
Not Completed | 11 | 8
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calmer Life | Enhanced Community Care | Total
Number analyzed (Participants) | 70 | 64 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.69 (9.394) | 67.14 (9.127) | 66.90 (9.235)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 48 | 109
  Male | 9 | 16 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 67 | 61 | 128
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 49 | 54 | 103
  White | 18 | 10 | 28
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70 | 64 | 134
Years of Education [Mean (Standard Deviation); unit: years] | 13.91 (2.853) | 13.28 (2.740) | 13.61 (2.807)
Marital Status [Count of Participants; unit: Participants]
  Married | 18 | 15 | 33
  Never Married | 7 | 11 | 18
  Separated | 3 | 2 | 5
  Divorced | 29 | 20 | 49
  Widowed | 13 | 16 | 29
Income [Count of Participants; unit: Participants]
  <$10,000 | 13 | 23 | 36
  $10,000 - $20,000 | 29 | 24 | 53
  $20,000 - $30,000 | 11 | 8 | 19
  $30,000 - $40,000 | 8 | 4 | 12
  $40,000 - $50,000 | 3 | 3 | 6
  $50,000 - $60,000 | 5 | 1 | 6
  ≥$60,000 | 1 | 1 | 2
Psychotropic Medication Use [Count of Participants; unit: Participants]
  Any psychotropic | 21 | 18 | 39
  Anti-anxiety | 7 | 7 | 14
  Anti-depressant | 16 | 13 | 29
  Anti-psychotic | 4 | 1 | 5
  Hypnotic/Sleep | 7 | 7 | 14
Medication Use, Total [Mean (Standard Deviation); unit: number of medications]
  Psychotropic | 0.50 (0.897) | 0.44 (0.778) | 0.47 (0.840)
  Non-psychotropic | 4.64 (3.323) | 4.51 (3.671) | 4.58 (3.480)
Diagnoses [Count of Participants; unit: Participants]
  None recorded | 5 | 4 | 9
  Generalized Anxiety Disorder (GAD) | 57 | 45 | 102
  Any Depressive Disorder | 35 | 34 | 69
  Post Traumatic Stress Dissorder (PTSD) | 5 | 3 | 8
  Social Phobia | 13 | 19 | 32
  Specific Phobia | 26 | 33 | 59
  Other Specificied Anxiety Disorder (OSAD) (GAD) | 4 | 10 | 14
  OSAD (Other) | 3 | 3 | 6
  Panic | 4 | 2 | 6
Service Use [Count of Participants; unit: Participants]
  Health Services | 64 | 56 | 120
  Hospital Admissions | 12 | 10 | 22
  Social Services | 22 | 17 | 39
  Psychological Services | 42 | 29 | 71
Expectancy Rating Scale (ERS) Cred [Mean (Standard Deviation); unit: units on a scale] — Measure of participant perception of the credibility of the intervention. Scores range from 3 to 30. Higher Scores indicate greater credibility. Population: The ERS was administered separately from other baseline measures, and not all participants were reached to complete this measure.
  units on a scale
    number analyzed (Participants) | 64 | 58 | 122
    (all) | 26.34 (4.213) | 25.03 (5.688) | 25.72 (4.991)
Expectancy Rating Scale (ERS) Exp [Mean (Standard Deviation); unit: units on a scale] — Measure of participant expectancy of improvement from intervention. Single item scores range from 0 to 10. Higher scores indicate greater expectations. Population: The ERS was administered separately from other baseline measures, and not all participants were reached to complete this measure.
  units on a scale
    number analyzed (Participants) | 64 | 58 | 122
    (all) | 8.58 (1.762) | 7.69 (2.650) | 8.16 (2.264)
Penn State Worry Questionnaire-A (PSWQ-A) [Mean (Standard Deviation); unit: units on a scale] — Brief measure of worry with 8 items measured on a 1-5 scale (1 = not at all typical, 3 = somewhat typical, 5 = very typical). Scores range from 8 to 40. Higher scores indicate greater anxiety.
  units on a scale | 26.73 (7.535) | 26.25 (6.933) | 26.50 (7.231)
Generalized Anxiety Disorder-7 (GAD-7) [Mean (Standard Deviation); unit: units on a scale] — Measure of Generalized Anxiety Disorder symptoms. 7 items rated from 0 (not at all) to 3 (nearly every day). Scores range from 0 to 21. Higher scores indicate greater GAD symptoms.
  units on a scale | 11.00 (5.421) | 10.56 (5.108) | 10.79 (5.259)
Geriatric Anxiety Inventory-SF (GAI-SF) [Mean (Standard Deviation); unit: units on a scale] — Five item scale with response options of yes = 1 and no = 0 to each item. Scores range from 0 to 5. Greater scores indicate greater anxiety.
  units on a scale | 3.39 (1.544) | 3.30 (1.752) | 3.34 (1.641)
Geriatric Depression Scale Short Form (GDS) [Mean (Standard Deviation); unit: units on a scale] — Brief measure of depression designed for use with older adults consisting of 15 items rated yes (1) or no (0). Scores range from 0 to 15. Higher scores indicate greater depression.
  units on a scale | 5.97 (3.547) | 5.61 (3.697) | 5.80 (3.610)
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: units on a scale] — Measure of sleep difficulties consisting of 7 items rated on a 0-4 scale. Scores range from 0 to 28. Higher scores indicate greater sleep difficulties.
  units on a scale | 13.44 (6.841) | 13.00 (6.264) | 13.23 (6.551)
Late-Life Function and Disability Instrument (LL-FDI) Disability Subscale - Frequency [Mean (Standard Deviation); unit: units on a scale] — Measure that assesses disability frequency across 16 life tasks and social roles. Frequencies for the 16 items are rated on a scale from 1 (never) to 5 (very often). Summary scores are transformed to scaled summary scores ranging from 0 to 100. Higher scores represent higher participation in tasks/higher functioning.
  units on a scale | 48.90 (6.281) | 48.05 (7.231) | 48.49 (6.739)
Late-Life Function and Disability Instrument (LL-FDI) Disability Subscale - Limitation [Mean (Standard Deviation); unit: units on a scale] — Measure that assesses disability limitations across 16 life tasks and social roles. Limitations for the 16 items are rated on a scale from 1 (completely limited) to 5 (not at all limited). Raw scores are transformed to scaled summary scores ranging from 0 to 100. Higher scores represent higher levels of capability of participating in tasks/higher functioning.
  units on a scale | 59.05 (10.799) | 59.38 (10.429) | 59.21 (10.585)
PTSD Checklist-5 (PCL-5) Total [Mean (Standard Deviation); unit: units on a scale] — Measure of PTSD symptoms. 20 items rated from 0 (not at all) to 4 (extremely). Scores range from 0 to 80. Higher scores = higher symptom severity.
  units on a scale | 28.77 (16.601) | 26.92 (16.157) | 27.89 (16.355)
Patient Health Questionnaire depression scale (PHQ 8) [Mean (Standard Deviation); unit: units on a scale] — Brief measure of depression symptoms consisting of 8 items rated from 0-3 (0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day). Scores range from 0 to 24. Higher scores indicate greater depression severity.
  units on a scale | 11.41 (6.076) | 11.13 (5.849) | 11.28 (5.948)
Brief RCOPE Positive Subscale [Mean (Standard Deviation); unit: units on a scale] — The Brief RCOPE is a 14 item measure of religious coping. The positive religious coping subscale includes 7 items rated from 0 (not at all) to 3 (great deal). Subscale scores range from 0-21. Higher scores indicate greater positive religious coping. Population: The Brief RCOPE was added to the study protocol after enrollment was underway, so data are not available for the full sample
  units on a scale
    number analyzed (Participants) | 58 | 55 | 113
    (all) | 24.22 (4.702) | 23.84 (4.144) | 24.04 (4.424)
Brief RCOPE Negative subscale [Mean (Standard Deviation); unit: units on a scale] — The Brief RCOPE is a 14 item measure of religious coping. The negative religious coping subscale includes 7 items rated from 0 (not at all) to 3 (great deal). Subscale scores range from 0-21. Higher scores indicate greater negative religious coping. Population: The Brief RCOPE was added to the study protocol after enrollment was underway, so data are not available for the full sample
  units on a scale
    number analyzed (Participants) | 58 | 55 | 113
    (all) | 10.38 (4.815) | 10.96 (5.044) | 10.66 (4.915)
Medical Outcomes Study 12-Item Short-Form Health Survey Physical Component Summary (SF-12 PCS) [Mean (Standard Deviation); unit: units on a scale] — Physical component summary score of the 12-item Medical Outcomes Study Short Form (SF-12), a measure of health-related quality of life. Summary raw scores are transformed to scale scores ranging from 0 to 100. Higher scores indicate higher levels of physical functioning.
  units on a scale | 38.38 (12.468) | 38.51 (11.498) | 38.44 (11.969)
Medical Outcomes Study 12-Item Short-Form Survey Mental Component Summary (SF-12 MCS) [Mean (Standard Deviation); unit: units on a scale] — Mental component summary score of the 12-item Medical Outcomes Study Short Form (SF-12), a measure of health-related quality of life. Summary raw scores are transformed to scale scores ranging from 0 to 100.Higher scores indicate higher levels of mental health functioning.
  units on a scale | 40.08 (9.708) | 40.14 (10.150) | 40.11 (9.884)

OUTCOME MEASURES:

1. Primary Outcome: Penn State Worry Questionnaire - A (PSWQ-A) at 6 Months
Description: Brief measure of worry with 8 items measured on a 1-5 scale (1 = not at all typical, 3 = somewhat typical, 5 = very typical). Scores range from 8 to 40. Higher scores indicate greater anxiety.
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 26.73 (7.53) | 26.25 (6.93)
  6 months | 22.04 (8.54) | 23.04 (7.17)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 6 month PSWQ-A, controlling for baseline PSWQ-A. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate of .05; Test type: Superiority; p = 0.77, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 0.08 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

2. Primary Outcome: Penn State Worry Questionnaire - A (PSWQ-A) at 9 Months
Description: as for outcome 1
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 26.73 (7.53) | 26.25 (6.93)
  9 months | 21.87 (8.72) | 20.18 (7.70)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 9 month PSWQ-A, controlling for baseline PSWQ-A. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.07, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 3.50 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

3. Primary Outcome: Generalized Anxiety Disorder-7 (GAD-7) at 6 Months
Description: Measure of Generalized Anxiety Disorder symptoms. 7 items rated from 0 (not at all) to 3 (nearly every day). Scores range from 0 to 21. Higher scores indicate greater GAD symptoms.
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 11.00 (5.42) | 10.56 (5.11)
  6 months | 7.13 (6.41) | 8.11 (5.69)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 6 month GAD-7, controlling for baseline GAD-7. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.34, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 0.92. (Numerator df = 1, Denominator df varies, as multiple imputation was used)

4. Primary Outcome: Generalized Anxiety Disorder-7 (GAD-7) at 9 Months
Description: as for outcome 3
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 11.00 (5.42) | 10.56 (5.11)
  9 months | 7.54 (5.51) | 6.62 (5.66)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 9 month GAD-7, controlling for baseline GAD-7. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.08, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 3.20 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

5. Secondary Outcome: Geriatric Anxiety Inventory - SF (GAI-SF) at 6 Months
Description: Five item scale with response options of yes = 1 and no = 0 to each item. Scores range from 0 to 5. Greater scores indicate greater anxiety.
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 3.39 (1.54) | 3.30 (1.75)
  6 months | 2.25 (2.00) | 2.48 (1.78)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 6 month GAI-SF, controlling for baseline GAI-SF. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.45, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 0.59 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

6. Secondary Outcome: Geriatric Anxiety Inventory - SF (GAI-SF) at 9 Months
Description: as for outcome 5
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 3.39 (1.54) | 3.30 (1.75)
  9 months | 2.65 (2.11) | 2.31 (1.71)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 9 month GAI-SF, controlling for baseline GAI-SF. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.13, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 2.37 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

7. Secondary Outcome: Patient Health Questionnaire Depression Scale (PHQ 8) at 6 Months
Description: Brief measure of depression symptoms consisting of 8 items rated from 0-3 (0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day). Scores range from 0 to 24. Higher scores indicate greater depression severity.
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 11.41 (6.08) | 11.13 (5.85)
  6 months | 7.28 (6.48) | 8.48 (6.06)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 6 month PHQ-8, controlling for baseline PHQ-8. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.52, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 0.42 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

8. Secondary Outcome: Patient Health Questionnaire Depression Scale (PHQ 8) at 9 Months
Description: as for outcome 7
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 11.41 (6.08) | 11.13 (5.85)
  9 months | 7.39 (6.35) | 7.00 (5.58)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 9 month PHQ-8, controlling for baseline PHQ-8. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.29, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 1.14 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

9. Secondary Outcome: Geriatric Depression Scale Short Form (GDS) at 6 Months
Description: Brief measure of depression designed for use with older adults consisting of 15 items rated yes (1) or no (0). Scores range from 0 to 15. Higher scores indicate greater depression.
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 5.97 (3.55) | 5.61 (3.70)
  6 months | 3.75 (3.42) | 4.33 (3.44)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 6 month GDS-SF, controlling for baseline GDS-SF. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.14, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 2.19 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

10. Secondary Outcome: Geriatric Depression Scale Short Form (GDS) at 9 Months
Description: as for outcome 9
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 5.97 (3.55) | 5.61 (3.70)
  9 months | 3.80 (3.49) | 3.92 (3.19)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 9 month GDS-SF, controlling for baseline GDS-SF. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.59, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 0.30 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

11. Secondary Outcome: Insomnia Severity Index (ISI) at 6 Months
Description: Measure of sleep difficulties consisting of 7 items rated on a 0-4 scale. Scores range from 0 to 28. Higher scores indicate greater sleep difficulties.
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 13.44 (6.84) | 13.00 (6.26)
  6 months | 10.08 (8.08) | 10.13 (7.16)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 6 month ISI, controlling for baseline ISI. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.64, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 0.22 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

12. Secondary Outcome: Insomnia Severity Index (ISI) at 9 Months
Description: as for outcome 11
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 13.44 (6.84) | 13.00 (6.26)
  9 months | 9.81 (7.65) | 9.51 (6.86)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 9 month ISI, controlling for baseline ISI. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.35, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 0.88 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

13. Secondary Outcome: Late-Life Function and Disability Instrument (LL-FDI) Disability Subscale - Frequency at 6 Months
Description: Measure that assesses disability frequency across 16 life tasks and social roles. Frequencies for the 16 items are rated on a scale from 1 (never) to 5 (very often). Summary scores are transformed to scaled summary scores ranging from 0 to 100. Higher scores represent higher participation in tasks/higher functioning.
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 48.90 (6.28) | 48.05 (7.23)
  6 months | 51.05 (7.30) | 49.83 (6.94)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 6 month LL-FDI, controlling for baseline LL-FDI. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.52, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 0.42 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

14. Secondary Outcome: Late-Life Function and Disability Instrument (LL-FDI) Disability Subscale - Frequency at 9 Months
Description: as for outcome 13
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 48.90 (6.28) | 48.05 (7.23)
  9 months | 50.85 (8.05) | 49.64 (8.97)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 9 month LL-FDI, controlling for baseline LL-FDI. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.92, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = .01(Numerator df = 1, Denominator df varies, as multiple imputation was used)

15. Secondary Outcome: Late-Life Function and Disability Instrument (LL-FDI) Disability Subscale - Limitation at 6 Months
Description: Measure that assesses disability limitations across 16 life tasks and social roles. Limitations for the 16 items are rated on a scale from 1 (completely limited) to 5 (not at all limited). Raw scores are transformed to scaled summary scores ranging from 0 to 100. Higher scores represent higher levels of capability of participating in tasks/higher functioning.
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 59.05 (10.80) | 59.39 (10.43)
  6 months | 64.54 (16.97) | 62.64 (13.30)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.59, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 0.29 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

16. Secondary Outcome: Late-Life Function and Disability Instrument (LL-FDI) Disability Subscale - Limitation
Description: as for outcome 15
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 59.05 (10.80) | 59.39 (10.43)
  9 months | 62.30 (13.86) | 62.45 (13.51)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.89, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 0.20 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

17. Secondary Outcome: Medical Outcomes Study 12-Item Short-Form Health Survey Physical Component Summary (SF-12 PCS) at 6 Months
Description: Physical component summary score of the 12-item Medical Outcomes Study Short Form (SF-12), a measure of health-related quality of life. Summary raw scores are transformed to scale scores ranging from 0 to 100. Higher scores indicate higher levels of physical functioning.
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 38.38 (12.47) | 38.51 (11.50)
  6 months | 37.86 (12.09) | 36.45 (11.95)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 6 month SF-12, controlling for baseline SF-12. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.64, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F= 0.23 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

18. Secondary Outcome: Medical Outcomes Study 12-Item Short-Form Health Survey Physical Component Summary (SF-12 PCS)
Description: as for outcome 17
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 38.38 (12.47) | 38.51 (11.50)
  9 months | 38.37 (13.26) | 36.93 (12.71)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 9 month SF-12, controlling for baseline SF-12. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.94, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 0.00 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

19. Secondary Outcome: Medical Outcomes Study 12-Item Short-Form Survey Mental Component Summary (SF-12 MCS) at 6 Months
Description: Mental component summary score of the 12-item Medical Outcomes Study Short Form (SF-12), a measure of health-related quality of life. Summary raw scores are transformed to scale scores ranging from 0 to 100.Higher scores indicate higher levels of mental health functioning.
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 40.08 (9.71) | 40.14 (10.15)
  6 months | 47.25 (12.17) | 45.91 (10.94)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.98, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 0.00 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

20. Secondary Outcome: Medical Outcomes Study 12-Item Short-Form Survey Mental Component Summary (SF-12 MCS) at 9 Months
Description: as for outcome 19
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 40.08 (9.71) | 40.14 (10.15)
  9 months | 46.98 (10.46) | 47.27 (11.57)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.88, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F= 0.02 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

21. Secondary Outcome: PTSD Checklist-5 (PCL-5) Total at 6 Months
Description: Measure of PTSD symptoms. 20 items rated from 0 (not at all) to 4 (extremely). Scores range from 0 to 80. Higher scores = higher symptom severity.
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 28.77 (16.60) | 18.02 (18.85)
  6 months | 26.92 (16.16) | 20.35 (16.11)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 6 month PCL-5, controlling for baseline PCL-5. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.31, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 1.02 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

22. Secondary Outcome: PTSD Checklist-5 (PCL-5) Total at 9 Months
Description: as for outcome 21
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
units on a scale
  Baseline | 28.77 (16.60) | 26.92 (16.16)
  9 months | 18.28 (17.39) | 18.53 (15.94)
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Analyses were ITT using PROC MI and PROC MI ANALYZE in conjunction with ANCOVA. We expected to reject the null hypothesis of no treatment group difference in 9 month PCL-5, controlling for baseline PCL-5. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.96, ANCOVA — P-value for treatment-group effect (CL vs ECC); Treatment group F = 0.00 (Numerator df = 1, Denominator df varies, as multiple imputation was used)

23. Secondary Outcome: Health Service Use at 6 Months
Description: Number of participants who had visited a health care provider (e.g., physician, nurse, physician's assistant) over the past 3 months.
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
Participants
  Baseline | 64 | 56
  6 months | 47 | 45
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; Test type: Superiority — We expected to reject the null hypothesis of no treatment group difference in 6 month health service use, controlling for baseline health service use. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; p = 0.52, Regression, Logistic — Parameter estimate for treatment group = 0.40 (SE = 0.63). Controlled for baseline health service use, ERS-expectancies and race/ethnicity; ITT analyses with PROC MI AND MI ANALYZE in conjunction with multiple logistic regression

24. Secondary Outcome: Health Service Use at 9 Months
Description: as for outcome 23
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
Participants
  Baseline | 64 | 56
  9 months | 52 | 39
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; We expected to reject the null hypothesis of no treatment group difference in 9 month health service use, controlling for baseline health service use. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.04, Regression, Logistic — Parameter estimate for treatment group = 1.79 (SE = 0.85). Controlled for baseline health service use, ERS-expectancies and race/ethnicity; ITT analyses with PROC MI AND MI ANALYZE in conjunction with multiple logistic regression

25. Secondary Outcome: Hospital Admissions at 6 Months
Description: Number of participants who were admitted to a hospital in the past 3 months.
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
Participants
  Baseline | 12 | 10
  6 months | 12 | 5
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; We expected to reject the null hypothesis of no treatment group difference in 6 month hospital admissions, controlling for baseline hospital admissions. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.04, Regression, Logistic — Parameter estimate for treatment group = 1.56 (SE = 0.74). Controlled for baseline health service use, ERS-expectancies and race/ethnicity; ITT analyses with PROC MI AND MI ANALYZE in conjunction with multiple logistic regression

26. Secondary Outcome: Hospital Admissions at 9 Months
Description: Number of participants who were admitted to a hospital in the past 3 months.
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
Participants
  Baseline | 12 | 10
  9 months | 14 | 3
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; We expected to reject the null hypothesis of no treatment group difference in 9 month hospital admissions, controlling for baseline hospital admissions. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.001, Regression, Logistic — Parameter estimate for treatment group = 2.96 (SE = 0.91). Controlled for baseline health service use, ERS-expectancies and race/ethnicity; ITT analyses with PROC MI AND MI ANALYZE in conjunction with multiple logistic regression

27. Secondary Outcome: Social Service or Resource Use at 6 Months
Description: Number of participants who received social services or resources over the past 3 months
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
Participants
  Baseline | 22 | 17
  6 months | 17 | 11
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; We expected to reject the null hypothesis of no treatment group difference in 6 month social service use, controlling for baseline social service use. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.42, Regression, Logistic — Parameter estimate for treatment group = 0.42 (SE = 0.51). Controlled for baseline health service use, ERS-expectancies and race/ethnicity; ITT analyses with PROC MI AND MI ANALYZE in conjunction with multiple logistic regression

28. Secondary Outcome: Social Service or Resource Use at 9 Months
Description: Number of participants who received social services or resources over the past 3 months
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
Participants
  Baseline | 22 | 17
  9 months | 18 | 14
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; We expected to reject the null hypothesis of no treatment group difference in 9 month social service use, controlling for baseline social service use. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.85, Regression, Logistic — Parameter estimate for treatment group = 0.09 (SE = 0.47). Controlled for baseline health service use, ERS-expectancies and race/ethnicity; ITT analyses with PROC MI AND MI ANALYZE in conjunction with multiple logistic regression

29. Secondary Outcome: Psychological Service Use at 6 Months
Description: Number of participants who discussed personal or emotional problems with a medical provider, clergy, mental health provider, or support group over the past 3 months
Time Frame: Baseline, 6 months
Population: 134 participants who completed baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
Participants
  Baseline | 42 | 29
  6 months | 31 | 31
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; We expected to reject the null hypothesis of no treatment group difference in 6 month psychological service use, controlling for baseline psychological service use. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.55, Regression, Logistic — Parameter estimate for treatment group = -0.28 (SE = 0.46). Controlled for baseline health service use, ERS-expectancies and race/ethnicity; ITT analyses with PROC MI AND MI ANALYZE in conjunction with multiple logistic regression

30. Secondary Outcome: Psychological Service Use at 9 Months
Description: as for outcome 29
Time Frame: Baseline, 9 months
Population: 134 participants who completed baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Calmer Life | Enhanced Community Care
Number analyzed (Participants) | 70 | 64
Participants
  Baseline | 42 | 29
  9 months | 26 | 20
Statistical Analysis 1: Comparison: Calmer Life vs Enhanced Community Care; We expected to reject the null hypothesis of no treatment group difference in 9 month psychological service use, controlling for baseline psychological service use. Race/ethnicity and ERS-expectancies significantly differed between groups at baseline and were included as covariates. A total of 134 participants allowed for 80% power to detect moderate group differences (d=.49) in primary and secondary outcomes given a 2-tailed type 1 error rate; Test type: Superiority; p = 0.54, Regression, Logistic — Parameter estimate for treatment group = -0.29 (SE = 0.47). Controlled for baseline health service use, ERS-expectancies and race/ethnicity; ITT analyses with PROC MI AND MI ANALYZE in conjunction with multiple logistic regression

ADVERSE EVENTS:
Time Frame: 2.5 years
Description: No adverse events were reported.
Arm/Group | Calmer Life | Enhanced Community Care
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/64
Other Adverse Events (participants affected / at risk) | 0/70 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT02391363/Prot_SAP_000.pdf